CLINICAL TRIAL: NCT06889389
Title: Effects of Pain Neuroscience Education and Therapeutic Exercise on Pain, Catastrophizing, Kinesiophobia and Upper Limb Function in Patients With Non-specific Neck Pain.
Brief Title: Effects of Education and Exercise on Pain, Psychosocial Factors, and Upper Limb Function in Non-specific Neck Pain.
Acronym: PNE-EXNP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Jaime Gascón Jaen, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI 90/2024; DPC.JGJ.241001 (Other: Miguel Hernández University)
Record Dates: First submitted 2025-03-05; First posted 2025-03-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain; Patient Education; Exercise Therapy; Fear; Pain
Keywords: Neck pain; Pain neuroscience education; Exercise therapy; Kinesiophobia; Pain catastrophizing
MeSH Terms: conditions — Neck Pain; Pain; Kinesiophobia | interventions — Educational Status; Exercise

STUDY DESIGN:
Intervention Model Description: This study follows a parallel-group design, where participants are randomly assigned to one of three intervention groups: (1) a control group receiving a placebo intervention (TENS device turned off, but participants are informed it is on at a very low, imperceptible intensity), (2) an exercise-only group, and (3) a group receiving both exercise and pain neuroscience education. The interventions are applied in a single session, and all groups undergo the same assessments before and after the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician will also be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education and Exercise group (Experimental): The investigator will proceed with pain neuroscience education focused on concepts related to movement-related fear and the benefits of exercise for 20 minutes. Specifically, the exercises presented in the generic part of the procedure will be discussed. To assess whether the education has produced changes in the subjects' beliefs, they will be reassessed regarding their beliefs about the exercises in relation to their neck pain following the education session. Subsequently, the subject will undergo the performance tests (Closed Kinetic Chain Upper Extremity Stability Test, Single Arm Military Press, and Seated Medicine Ball Throw), which will be carried out by a second investigator. The exercise intervention will then proceed using variations of the performance tests, also conducted by the second investigator. Specifically, the load or execution time will be increased until the participant reports a perceived fatigue of 4-6 (moderate to strong) on the modified Borg scale.
  Interventions: Behavioral: Education; Other: Excercise
- Exercise group (Experimental): This group does not include pain neuroscience education. Following the initial assessment, the subject will be left alone for 20 minutes with instructions to think about the exercises but not to perform them. Subsequently, the subject will undergo the performance tests (Closed Kinetic Chain Upper Extremity Stability Test, Single Arm Military Press, and Seated Medicine Ball Throw), which will be carried out by a second investigator. The exercise intervention will then proceed using variations of the performance tests, also conducted by the second investigator. Specifically, the load or execution time will be increased until the participant reports a perceived fatigue of 4-6 (moderate to strong) on the modified Borg scale.
  Interventions: Other: Excercise
- Control group (Placebo Comparator): This group does not include pain neuroscience education or exercise. Following the initial assessment, the subject will be left alone for 20 minutes with instructions to think about the exercises but not to perform them. Subsequently, subjects in this group will receive a placebo intervention. A TENS device will be placed on them and kept turned off for 15 minutes. Subjects will be informed that the device is working at a very low intensity, too weak to be perceived. Additionally, performance tests will not be assessed in this group.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Education — The intervention consists of 20 minutes of pain neuroscience education, focused on concepts related to movement-related fear and the benefits of exercise for managing pain. Specific exercises, mentioned in the generic part of the procedure, will be discussed during this session. This intervention aims to modify the subjects' beliefs regarding exercises and their neck pain.
  Other Names: Pain Neuroscience Education; Pain Education Therapy
  Arms: Education and Exercise group
Other: Excercise — The exercise intervention includes performance tests and variations of these tests used as exercises, such as the Closed Kinetic Chain Upper Extremity Stability Test, Single Arm Military Press, and Seated Medicine Ball Throw. Variations of these performance tests will be implemented, with adjustments made to the load or execution time until the participant reports a perceived fatigue of 4-6 (moderate to strong) on the modified Borg scale.
  Other Names: Physical exercise; Physical activity
  Arms: Education and Exercise group; Exercise group
Other: Placebo — The placebo intervention involves the application of a TENS device, which will be placed on the participant and kept turned off for 15 minutes. Subjects will be informed that the device is working at a very low intensity, too weak to be perceived. This intervention aims to simulate the experience of treatment without delivering any therapeutic effect.
  Arms: Control group

SUMMARY:
Pain neuroscience education is currently one of the techniques being explored in physiotherapy for pain management. The benefits of this technique are gradually becoming evident in various published studies. So far, it has been widely studied for its short-term effects, but the education provided has typically been generic, not focused on exercise. However, it is suggested that this technique should be combined with exercise to achieve the expected outcomes. Therefore, pain education should be tailored to the specific physical activities the subject will perform to maximise its effectiveness. The primary aim of this study is to analyse the outcome of combining exercise with tailored pain neuroscience education on aspects such as pain, kinesiophobia, catastrophizing, exercise conceptualization, and upper limb function in subjects with neck pain. The secondary aim is to evaluate the relationship between kinesiophobia and catastrophizing and their impact on the results of various upper limb performance tests. Finally, the effects of therapeutic exercise alone will be compared with those of therapeutic exercise combined with pain neuroscience education, focusing on pain, kinesiophobia, catastrophizing, and exercise conceptualization. A double-blind, randomised clinical trial has been designed, in which three intervention protocols will be applied to 81 subjects with non-specific neck pain: education with exercise, exercise alone, and placebo alone. Subjects with non-specific neck pain who meet the inclusion criteria will be enrolled. Demographic characteristics of the subjects, as well as pain, kinesiophobia, catastrophizing, and upper limb performance test scores, will be assessed. This study aims to explore the potential relevance of a pain neuroscience education session prior to therapeutic exercise, as well as to influence the clinical recommendations made by clinicians during treatment.

DETAILED DESCRIPTION:
In recent years, education in pain neuroscience has been shown to have a positive impact on pain subjects. However, the education provided is often generic and not adapted to exercise, although it is recommended that this therapy should be combined with exercise. Therefore, the aim of this study is to assess the results of the combination of exercise and pain neuroscience education focused on the exercise to be performed by subjects in pain or kinesiophobia. Therefore, the main objective of the study is to evaluate the effects of pain neuroscience education in non-specific neck pain on pain intensity, kinesiophobia, catastrophizing, exercise conceptualization and upper limb functionality itself in subjects with non-specific neck pain. The specific objective is to compare the effect of therapeutic exercise alone with the effect of therapeutic exercise in combination with pain neuroscience education on pain, kinesiophobia, catastrophizing and exercise conceptualization. Similarly, the aim is to determine the relationship between kinesiophobia and catastrophism and the results obtained in upper limb performance tests. For this purpose, the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), the Seated Medicine Ball Throw test (SMBT) and the Single Arm Military Press (SAMP) have been chosen, the first two of which have not been studied in patients with non-specific neck pain to date. This study aims to have an impact on the possible relevance of a pain neuroscience education session prior to therapeutic exercise, as well as on the clinical recommendations made by healthcare professionals during treatment.

DESIGN The study consists of a randomised, double-blind clinical trial. Subjects will be randomised into 3 groups: control group, where subjects will receive a placebo (TENS off, in this case); intervention group 1, where pain neuroscience education (PNE) and exercise will be applied; and intervention group 2, to which only exercise will be applied. The allocation will be blinded to the subject and to one of the two investigators. SELECTION CRITERIA Inclusion criteria: o Adults aged between 18 and 65 years. o Subjects with non-specific neck pain at the time of the intervention reaching at least a 3 on the Numerical Pain Rating Scale (NPRS scale). Exclusion criteria: o Pregnancy o Severe illnesses: diabetes, cancer, neurological, depression, etc... o Cognitive disorders or illnesses. o Subjects who have received physiotherapy treatment in the last month. o Subjects who are receiving concomitant physiotherapy treatment for this pathology. o Subjects with specific neck pain, such as any traumatic pathology, whiplash or with a diagnosis associated with neurological compromise or peripheral nerve damage. o Physiotherapy students or professional physiotherapists. Subjects included in the study must complete the informed consent form, meet the inclusion criteria and not meet the exclusion criteria. Prior to any type of procedure, subjects will be informed about the study and about their right to discontinue their participation and/or request the withdrawal of their data at any time.

DESCRIPTION OF THE PROCEDURE At the beginning, all subjects will sign the informed consent form, demographic data will be recorded by means of an interview and a questionnaire specifically designed for the work. After that, baseline measurements of outcome variables will be taken. Fear of movement and kinesiophobia will be measured with the Tampa Scale of Kinesiophobia (TSK- 11SV), pain catastrophizing with the Pain and Catastrophizing Scale (PCS), and subject's beliefs about pain with the Pain Beliefs Questionnaire (PBQ). The Spanish validated versions of all the aforementioned scales will be used. The Numerical Pain Rating Scale (NPRS) will be used to assess subjects' current pain and spontaneous or evoked pain intensity. Researcher A will then show each subject images of the 3 performance tests they will have to perform, as well as provide an explanation of their execution: Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), Single Arm Military Press (SAMP) and Seated Medicine Ball Throw Test (SMBT). Regardless of whether subjects are later assigned to the exercise group or not. These tests are among the most widely used tests to measure upper limb function, although they have not been studied in subjects with non-specific neck pain. The Single Arm Military Press (SAMP) test is the only performance-based measure of upper limb disability that was designed specifically for subjects with neck pain. All these tests involve active movements that could be conditioned by the subject's pain and beliefs related to kinesiophobia, so they could be of great use to observe whether an educational approach decreases upper limb dysfunction. Finally, subjects' beliefs about the exercises explained in relation to their pathology will be assessed by means of a questionnaire specifically designed for this purpose. After this procedure is completed by all participants, they will be randomised into three groups, using a randomisation website (Research Randomizer, n.d.) and will undergo a physiotherapy session that includes different approaches for each group.

In the PNE and exercise group the investigator will proceed with pain neuroscience education focused on concepts related to movement-related fear and the benefits of exercise for 20 minutes. Specifically, the exercises presented in the generic part of the procedure will be discussed. To assess whether the education has resulted in changes to the subjects' beliefs, they will be reassessed regarding their beliefs about the exercises in relation to their neck pain following the education session. Afterward, subjects will complete psychosocial scales and rate their pain and evoked pain at that moment independently, without the need for the researcher to be present, in order to ensure blinding. Subsequently, the subject will undergo the performance tests in a randomised order (Closed Kinetic Chain Upper Extremity Stability Test, Single Arm Military Press, and Seated Medicine Ball Throw), which will be conducted by a second investigator who is unaware of whether the subject has received education. The exercise intervention will then proceed using variations of the performance tests, also carried out by the second investigator. Specifically, the load or execution time will be increased until the participant reports a perceived fatigue of 4-6 (moderate to strong) on the modified Borg scale. Finally, the participant will autonomously complete the scales, rate their pain and exercise-related questions for the final time.

The exercise group does not include pain neuroscience education. Following the initial assessment, the subject will be left alone for 20 minutes with instructions to think about the exercises but not to perform them. Afterward, subjects will complete psychosocial scales and will rate their pain and evoked pain at that moment independently, without the need for the researcher to be present, in order to ensure blinding. Subsequently, the subject will undergo the performance tests in a randomised order (Closed Kinetic Chain Upper Extremity Stability Test, Single Arm Military Press, and Seated Medicine Ball Throw), which will be conducted by a second investigator who is unaware of whether the subject has received education. The exercise intervention will then proceed using variations of the performance tests, also carried out by the second investigator. Specifically, the load or execution time will be increased until the participant reports a perceived fatigue of 4-6 (moderate to strong) on the modified Borg scale. Finally, the participant will independently complete the scales, rate their pain, evoked pain, and exercise-related questions one final time.

The control group does not receive pain neuroscience education or exercise. Following the initial assessment, the subject will be left alone for 20 minutes with instructions to think about the exercises but not to perform them. Afterward, subjects will independently complete psychosocial scales and will rate their pain and evoked pain at that moment, without the need for the researcher to be present, in order to ensure blinding. Subsequently, participants in this group will receive a placebo intervention administered by a second investigator. A TENS device will be placed on them and kept turned off for 15 minutes. subjects will be informed that the device is operating at a very low intensity, too weak to be perceived. Additionally, performance tests will not be assessed in this group. Finally, the participant will autonomously complete the scales, rate their pain and exercise-related questions for the final time. Therefore, all groups will be assessed 3 times during the session. The first time they will be accompanied by the first investigator, who will answer any questions that may arise. The second and third time the subject will do it autonomously, unaccompanied by any researcher, to avoid bias.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 65 years
* Subjects with non-specific neck pain at the time of the intervention, scoring at least 3 on the NPRS scale.

Exclusion Criteria:

* Pregnancy
* Severe illnesses: diabetes, cancer, neurological conditions, depression, etc.
* Subjects impairments or disorders
* Subjects who have received physiotherapy treatment within the last month
* Subjects currently undergoing concurrent physiotherapy treatment for this condition
* Subjects with specific neck pain, such as any traumatic pathology, whiplash, or diagnoses associated with neurological compromise or peripheral nerve damage
* Physiotherapy students or professional physiotherapists

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Kinesiophobia Level from Baseline to the End of the Interventions as Assessed by the Tampa Scale for Kinesiophobia (TSK-11SV) | Baseline (Day 1), post-education/rest (Day 1), and post-intervention (Day 1).
  The level of kinesiophobia will be assessed using the Tampa Scale for Kinesiophobia (TSK-11SV). This scale evaluates kinesiophobia (fear of movement) through 11 statements, which participants must rate on a Likert scale from 1 to 4, where 1 indicates strongly disagree and 4 indicates strongly agree. Higher scores reflect greater kinesiophobia (minimum score: 11; maximum score: 44). The validated Spanish version of the scale will be used.
Change in Pain Beliefs from Baseline to the End of the Interventions as Assessed by the Pain Beliefs Questionnaire (PBQ). | Baseline (Day 1), post-education/rest (Day 1), and post-intervention (Day 1).
  Pain beliefs will be assessed using the Pain Beliefs Questionnaire (PBQ), which evaluates beliefs regarding the causes, consequences, and necessary treatment of pain. The questionnaire is divided into two subscales: "organic" and "psychological." It consists of 12 items, with 8 items belonging to the "organic" subscale and 4 to the "psychological" subscale. The PBQ uses a 6-point Likert scale ranging from "Always" to "Never," corresponding to scores of 6 and 1, respectively. Higher scores on each subscale indicate that the respondent considers the corresponding pain-related beliefs to be of greater importance.
Change in Catastrophizing Level from Baseline to the End of the Interventions as Assessed by the Pain and Catastrophizing Scale (PCS). | Baseline (Day 1), post-education/rest (Day 1), and post-intervention (Day 1).
  The level of catastrophizing will be assessed using the Pain and Catastrophizing Scale (PCS). This scale evaluates catastrophizing in response to pain and the negative and exaggerated perception of the painful experience. It consists of 13 statements describing different thoughts and feelings that may be associated with pain. The participant is required to indicate the extent to which they experience these thoughts and feelings when they are in pain. Each statement is rated on a Likert scale from 0 to 4, where 0 means "not at all" and 4 means "all the time." Higher scores indicate a higher degree of catastrophizing. The validated Spanish version of the scale will be used.
Change in Pain Intensity from Baseline to the End of the Interventions as Assessed by the Numerical Pain Rating Scale (NPRS). | Baseline (Day 1), post-education/rest (Day 1), and post-intervention (Day 1).
  Pain intensity will be assessed using the Numerical Pain Rating Scale (NPRS). This scale evaluates the intensity of pain experienced by the participant, using a 10-point scale, where 0 represents no pain and 10 represents the maximum possible pain. Higher scores correspond to greater pain intensity.
Change in Evoked Pain Intensity from Baseline to the End of the Interventions as Assessed by the Numerical Pain Rating Scale (NPRS) | Baseline (Day 1), post-education/rest (Day 1), and post-intervention (Day 1).
  Evoked pain will be assessed using the Numerical Pain Rating Scale (NPRS). Participants will be asked to perform a movement that evokes pain related to their condition. Pain intensity will then be evaluated on a 10-point scale, where 0 represents no pain and 10 represents the maximum possible pain. Higher scores correspond to greater pain intensity.

SECONDARY OUTCOMES:
Demographic data | Baseline (Day 1).
  Participants will complete a demographic questionnaire, including descriptive variables such as age, sex, weight, height, level of physical activity, comorbidities, duration of pain, side of pain, and smoking status.
Change in Beliefs About Specific Exercises from Baseline to the End of the Interventions as Assessed by the Custom Questionnaire on Beliefs About Specific Exercises. | Baseline (Day 1), post-education/rest (Day 1), and post-intervention (Day 1).
  Beliefs about specific exercises in relation to pain will be assessed using a custom questionnaire. The questionnaire evaluates the participants' beliefs regarding the specific exercises they will perform. Participants will first be shown photographs of the exercises they are required to do, and then they will respond to the questionnaire by selecting a number on a visual analogue scale from 1 to 10, where 1 indicates "strongly disagree" and 10 indicates "strongly agree." Higher scores reflect stronger beliefs about the exercises in relation to their pain.
  This questionnaire was specifically designed for this study and is being used for data collection.
Average pain intensity over the last 7 days as assessed by the numerical pain rating scale (NPRS) | Baseline (Day 1).
  Average pain intensity over the last 7 days will be assessed using the Numerical Pain Rating Scale (NPRS). This scale evaluates both the average pain intensity experienced by the participant over the last 7 days, using a 10-point scale where 0 represents no pain and 10 represents the maximum possible pain. Higher scores correspond to greater pain intensity.
Worst Pain Intensity in the Last 7 Days as Assessed by the Numerical Pain Rating Scale (NPRS) | Baseline (Day 1).
  The worst pain intensity over the last 7 days will be assessed using the Numerical Pain Rating Scale (NPRS). This scale evaluates the worst pain intensity experienced by the participant over the past 7 days, using a 10-point scale where 0 represents no pain and 10 represents the maximum possible pain. Higher scores indicate greater pain intensity.
Functional Performance of the Upper Extremity as Assessed by the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) | Post-education/rest (Day 1).
  Functional performance of the upper extremities will be assessed using the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), a test designed to evaluate upper limb stability and control. During the test, male participants will adopt a push-up position, while female participants will assume a modified push-up position (knees on the ground). Both hands will be placed on two strips on the floor at the same height, with a distance of 91.4 cm between them. In these positions, participants will be required to move one hand to touch the back of the opposite hand, then return to the starting position, repeating the movement with the other hand, for 15 seconds. The test will be performed for three 15-second repetitions at maximum effort, with a 45-second rest between each repetition. The outcome measure will be the average number of touches (mean of the number of touches from the three attempts).
Functional Performance of the Upper Extremity as Assessed by the Single Arm Military Press test (SAMP test) | Post-education/rest (Day 1).
  Functional performance of the upper extremity will be assessed using the Single Arm Military Press (SAMP). This performance-based measure is designed to assess upper extremity strength during an overhead activity, aimed at differentiating between healthy individuals and those with varying levels of nonspecific neck pain and upper extremity disability. The exercise is performed with participants standing, with their feet shoulder-width apart, holding a 1 kg dumbbell at shoulder height with their dominant hand. Participants are instructed to lift the dumbbell overhead, performing a full shoulder flexion and elbow extension. The test consists of repeating this motion as quickly as possible for 30 seconds with maximal effort. The SAMP score is determined by counting the number of correct repetitions completed in 30 seconds. The test is stopped if the participant is unable to complete another correct repetition.
Functional Performance of the Upper Extremities as Assessed by the Seated Medicine Ball Throw Test (SMBT) | Post-education/rest (Day 1).
  Functional performance of the upper extremities will be assessed using the Seated Medicine Ball Throw Test (SMBT). Participants will sit with their back against the wall, legs extended, holding a 2 kg medicine ball with arms at 90° shoulder abduction and elbows flexed at chest height. They will throw the ball forward as far as possible without losing contact with the wall. The distance will be measured by a tape placed 10 meters from the subject's starting point. Three maximum effort throws will be performed with 1-minute rests between each, and the result will be the average of the three throws.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica de Franscisco Ortega Rehabilitación Avanzada S.L., Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control. Man Ther. 2008 Feb;13(1):2-11. doi: 10.1016/j.math.2007.06.003. Epub 2007 Aug 16. PMID 17702636
- [Background] Thompson DP, Urmston M, Oldham JA, Woby SR. The association between cognitive factors, pain and disability in patients with idiopathic chronic neck pain. Disabil Rehabil. 2010;32(21):1758-67. doi: 10.3109/09638281003734342. PMID 20350122
- [Background] Stagg NJ, Mata HP, Ibrahim MM, Henriksen EJ, Porreca F, Vanderah TW, Philip Malan T Jr. Regular exercise reverses sensory hypersensitivity in a rat neuropathic pain model: role of endogenous opioids. Anesthesiology. 2011 Apr;114(4):940-8. doi: 10.1097/ALN.0b013e318210f880. PMID 21386701
- [Background] Sluka KA, Frey-Law L, Hoeger Bement M. Exercise-induced pain and analgesia? Underlying mechanisms and clinical translation. Pain. 2018 Sep;159 Suppl 1(Suppl 1):S91-S97. doi: 10.1097/j.pain.0000000000001235. PMID 30113953
- [Background] Senarath ID, Chen KK, Weerasekara I, de Zoete RMJ. Exercise-induced hypoalgesic effects of different types of physical exercise in individuals with neck pain: A systematic review and meta-analysis. Pain Pract. 2023 Jan;23(1):110-122. doi: 10.1111/papr.13150. Epub 2022 Aug 2. PMID 35869789
- [Background] Osborn W, Jull G. Patients with non-specific neck disorders commonly report upper limb disability. Man Ther. 2013 Dec;18(6):492-7. doi: 10.1016/j.math.2013.05.004. Epub 2013 May 29. PMID 23726285
- [Background] Ortego G, Villafane JH, Domenech-Garcia V, Berjano P, Bertozzi L, Herrero P. Is there a relationship between psychological stress or anxiety and chronic nonspecific neck-arm pain in adults? A systematic review and meta-analysis. J Psychosom Res. 2016 Nov;90:70-81. doi: 10.1016/j.jpsychores.2016.09.006. Epub 2016 Sep 9. PMID 27772562
- [Background] Luque-Suarez A, Martinez-Calderon J, Falla D. Role of kinesiophobia on pain, disability and quality of life in people suffering from chronic musculoskeletal pain: a systematic review. Br J Sports Med. 2019 May;53(9):554-559. doi: 10.1136/bjsports-2017-098673. Epub 2018 Apr 17. PMID 29666064
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Lee DR, Kim LJ. Reliability and validity of the closed kinetic chain upper extremity stability test. J Phys Ther Sci. 2015 Apr;27(4):1071-3. doi: 10.1589/jpts.27.1071. Epub 2015 Apr 30. PMID 25995559
- [Background] Javdaneh N, Saeterbakken AH, Shams A, Barati AH. Pain Neuroscience Education Combined with Therapeutic Exercises Provides Added Benefit in the Treatment of Chronic Neck Pain. Int J Environ Res Public Health. 2021 Aug 22;18(16):8848. doi: 10.3390/ijerph18168848. PMID 34444594
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Background] Dzakpasu FQS, Carver A, Brakenridge CJ, Cicuttini F, Urquhart DM, Owen N, Dunstan DW. Musculoskeletal pain and sedentary behaviour in occupational and non-occupational settings: a systematic review with meta-analysis. Int J Behav Nutr Phys Act. 2021 Dec 13;18(1):159. doi: 10.1186/s12966-021-01191-y. PMID 34895248
- [Background] Decleve P, Van Cant J, De Buck E, Van Doren J, Verkouille J, Cools AM. The Self-Assessment Corner for Shoulder Strength: Reliability, Validity, and Correlations With Upper Extremity Physical Performance Tests. J Athl Train. 2020 Apr;55(4):350-358. doi: 10.4085/1062-6050-471-18. Epub 2020 Feb 13. PMID 32053404
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Clarke CL, Ryan CG, Martin DJ. Pain neurophysiology education for the management of individuals with chronic low back pain: systematic review and meta-analysis. Man Ther. 2011 Dec;16(6):544-9. doi: 10.1016/j.math.2011.05.003. Epub 2011 Jun 25. PMID 21705261
- [Background] Bushnell MC, Ceko M, Low LA. Cognitive and emotional control of pain and its disruption in chronic pain. Nat Rev Neurosci. 2013 Jul;14(7):502-11. doi: 10.1038/nrn3516. Epub 2013 May 30. PMID 23719569
- [Background] Borms D, Maenhout A, Cools AM. Upper Quadrant Field Tests and Isokinetic Upper Limb Strength in Overhead Athletes. J Athl Train. 2016 Oct;51(10):789-796. doi: 10.4085/1062-6050-51.12.06. Epub 2016 Nov 11. PMID 27834503
- [Background] Cibulka MT, White DM, Woehrle J, Harris-Hayes M, Enseki K, Fagerson TL, Slover J, Godges JJ. Hip pain and mobility deficits--hip osteoarthritis: clinical practice guidelines linked to the international classification of functioning, disability, and health from the orthopaedic section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2009 Apr;39(4):A1-25. doi: 10.2519/jospt.2009.0301. No abstract available. PMID 19352008
- [Background] Bier JD, Scholten-Peeters WGM, Staal JB, Pool J, van Tulder MW, Beekman E, Knoop J, Meerhoff G, Verhagen AP. Clinical Practice Guideline for Physical Therapy Assessment and Treatment in Patients With Nonspecific Neck Pain. Phys Ther. 2018 Mar 1;98(3):162-171. doi: 10.1093/ptj/pzx118. PMID 29228289
- [Background] Beltran-Alacreu H, Lopez-de-Uralde-Villanueva I, Fernandez-Carnero J, La Touche R. Manual Therapy, Therapeutic Patient Education, and Therapeutic Exercise, an Effective Multimodal Treatment of Nonspecific Chronic Neck Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2015 Oct;94(10 Suppl 1):887-97. doi: 10.1097/PHM.0000000000000293. PMID 25888653
- [Background] Alreni ASE, Aboalmaty HRA, De Hertogh W, Wakwak OSM, McLean SM. Construct validity of the Single Arm Military Press (SAMP) test for upper limb function in patients with neck pain. Musculoskelet Sci Pract. 2023 Feb;63:102707. doi: 10.1016/j.msksp.2022.102707. Epub 2022 Dec 7. PMID 36525941

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT06889389/Prot_SAP_002.pdf
  • Informed Consent Form (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT06889389/ICF_003.pdf